CLINICAL TRIAL: NCT05180708
Title: A Multicenter, Phase 3 Randomized, Double-Blind, Vehicle-controlled Study Evaluating the Safety and Efficacy of QTORIN 3.9% Rapamycin Anhydrous Gel in the Treatment of Pachyonychia Congenita
Acronym: VAPAUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Palvella Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PALV-05
Record Dates: First submitted 2021-12-20; First posted 2022-01-06 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Pachyonychia Congenita
MeSH Terms: conditions — Pachyonychia Congenita

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator)
  Interventions: Drug: QTORIN 3.9% rapamycin anhydrous gel
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: QTORIN 3.9% rapamycin anhydrous gel — QTORIN 3.9% rapamycin anhydrous gel
  Arms: Active
Drug: Vehicle — Matching vehicle (QTORIN anyhydrous gel)
  Arms: Vehicle

SUMMARY:
This study evaluates the safety and efficacy of QTORIN 3.9% rapamycin anhydrous gel in the treatment of adults with Pachyonychia Congenita. This study includes a screening period, baseline period and 6-month treatment period.

ELIGIBILITY:
Key Inclusion Criteria:

* Adult patients, 18 years or older (16 years or older in the UK)
* Diagnosed with Pachyonychia Congenita (PC), genetically confirmed

Key Exclusion Criteria:

* Any history of allergy or hypersensitivity to sirolimus, or sirolimus-like medications.
* Any significant concurrent condition (including conditions involving or inferior to the ankle) that could adversely affect the patient's participation and/or the assessment of the safety and efficacy in the study.
* Participation in any other interventional clinical research trial within 30 days prior to the screening visit or during the patient's participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Patient Global Assessment of Activities Difficulty Scale | 6 months

SECONDARY OUTCOMES:
Pain at its worst as assessed by numerical rating scale | 6 months
PROMIS physical function | 6 months
Patient global impression of severity (PGI-S) | 6 months
Patient global impression of change (PGI-C) | 6 months
Clinician global impression of severity (CGI-S) | 6 months
Clinician global impression of change (CGI-C) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Amy Paller, MD, Study Chair — Northwestern University; Joyce Teng, MD, Principal Investigator — Stanford University; David Hansen, MD, Principal Investigator — University of Utah
Locations (8):
- United States (7):
  - Stanford University, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Park Avenue Dermatology, Orange Park, Florida
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Oregon Health and Sciences University, Portland, Oregon
  - DermResearch, Inc., Austin, Texas
  - University of Utah, Murray, Utah
- Royal London Hospital, London, Whitechapel, United Kingdom

REFERENCES:
- See also: PC Project — http://www.pachyonychia.org/
- See also: Palvella Therapeutics, Inc. — http://palvellatx.com